CLINICAL TRIAL: NCT05343169
Title: Evaluation of a Community-based Education, Navigation, and Support (CENS) Intervention to Reduce Opioid-related Harms Among Military Veterans
Brief Title: Community-based Education, Navigation, and Support Intervention for Military Veterans
Acronym: CENS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA052426 (NIH)
Record Dates: First submitted 2022-03-08; First posted 2022-04-25 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Overdose; Opioid Use Disorder; HIV Infections
MeSH Terms: conditions — Drug Overdose; Opioid-Related Disorders; HIV Infections | interventions — Therapeutics; Self Care; Educational Status; Social Work; Palliative Care

STUDY DESIGN:
Intervention Model Description: Two arm, parallel randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CENS Intervention (Experimental): Peer outreach workers will deliver Overdose Education and Naloxone to participants and provide education, navigation, and support during the 9-month intervention
  Interventions: Behavioral: Overdose Education and Naloxone Distribution; Behavioral: Advanced Education in Safer Substance Use, Treatment, and Self-Care; Behavioral: Social Service and Health Navigation; Behavioral: Peer Social Support
- Control (Other): Participants will receive Overdose Education and Naloxone and referrals to treatment
  Interventions: Behavioral: Overdose Education and Naloxone Distribution

INTERVENTIONS:
Behavioral: Overdose Education and Naloxone Distribution — Education on OD risk behaviors and methods for responding to an OD, including naloxone use.
  Duration and dose: Single 20-minute training at time of enrollment, provided to all participants in both arms
  Other Names: OEND
Behavioral: Advanced Education in Safer Substance Use, Treatment, and Self-Care — Education about misinformation about OAT, self-care, SEP services, HIV/HCV treatment Duration/dose: 9 mos., monthly ~2 hr. group sessions + ongoing access to video archive of recorded trainings.
  Other Names: Education
  Arms: CENS Intervention
Behavioral: Social Service and Health Navigation — Help navigate access and barriers to healthcare, motivation and health goals Duration/dose: 9 mos., monthly face-to-face sessions to set goals and schedule appts, phone calls between sessions > 1x/wk.
  Other Names: Navigation
  Arms: CENS Intervention
Behavioral: Peer Social Support — Support with social (re)integration, isolation, relationship building Duration/dose: 9 mos., monthly face-to-face events and phone calls/texts between sessions > 1x/wk.
  Other Names: Support
  Arms: CENS Intervention

SUMMARY:
Military veterans in the U.S. represent one of the populations most disproportionately impacted by the current opioid crisis. Veterans who use opioids and are not connected to the VA healthcare system have high rates of homelessness and experience higher prevalence of comorbid substance use disorder and mental health diagnoses than their "service-connected" counterparts. Due to these vulnerabilities and the observed barriers to testing and treatment among veterans-especially substance- and mental health-related stigma, drug naiveté, and limited support networks-veterans who use opioids represent a critical target for interventions designed to mitigate overdose and HIV/HCV risk behaviors. For socially isolated veterans and veterans with limited access to healthcare, programs that work outside of formal healthcare institutions and agencies are desperately needed. This application proposes to achieve the following Aims: 1) Evaluate the effectiveness of a peer-delivered, community-based education, navigation and support (CENS) intervention to reduce opioid-related risk behaviors; 2) Examine factors that mediate (e.g., knowledge, self-efficacy, self-stigma) and moderate (e.g., mental health, pain/OUD severity, age) intervention effectiveness; and 3) Explore intervention participants' and peer outreach staff perspectives on implementation as well as barriers to and facilitators of intervention effectiveness. The proposed intervention will be delivered by veteran peer outreach workers. The study will recruit 300 veterans with opioid use disorder to participate in a randomized controlled trial. The CENS intervention will engage 150 participants in ongoing educational sessions, healthcare and treatment navigation, and social support (involving both one-on-one and group social integration protocols) designed to improve self-efficacy, reduce self-stigma, increase service and healthcare utilization, and bolster knowledge. This study stands to contribute a timely, culturally-tailored innovation to overdose and HIV/HCV prevention-as-usual that, informed by the theory of triadic influence, directly confronts the social, intrapersonal, and structural-level barriers to opioid-related risk reduction among veterans. Study findings will be of great interest to community-based and civic healthcare organizations that provide overdose and HIV/HCV risk reduction outreach, as well as to agencies committed to improving healthcare engagement among veterans.

DETAILED DESCRIPTION:
The U.S. remains in a public health crisis involving opioid-related morbidity and mortality,1 and military veterans have been disproportionately impacted. Among veterans who use VA hospitals, the prevalence of OD deaths from non-synthetic opioids roughly doubled between 2001 and 2009, and deaths among this population have continued to rise dramatically, showing a 65 percent increase from 2010 to 2016 alone. This trend is grounded in high rates of concurrent prescription opioid (PO) and benzodiazepine use, but transitions from POs to heroin9 have been a recent driver of OD mortality and the disproportionately high HIV and HCV infection rates among veterans.1 Additionally, much of the scientific knowledge about health risks among veterans who use opioids (VWUO) comes from VA samples, which represent less than half of all military veterans. Veterans who do not have VA access or choose not to use it, include many of those most historically disadvantaged and at greatest risk of opioid-related harm. Rates of 'other than honorable' discharges for active duty personnel with alcohol or substance use issues have increased, excluding them from VA care and resulting in underestimates of opioid-related harms among the broader veteran population. For example, the prevalence of HCV infection-driven primarily by injection drug use-has been estimated at 11-18% among veterans who utilize the VA but up to 45% among the sizable population of homeless veterans, most of whom do not. Irrespective of benefit status, many veterans with substance and alcohol use disorders avoid substance use treatment, healthcare, and supported social services, such as opioid agonist therapy, housing and employment assistance, syringe service programs, mental health treatment, and HIV/HCV testing and treatment. Social isolation and a sense of alienation from civilian society have long represented important barriers to working with veteran populations and highlight the need for targeted, culturally sensitive interventions that reach at-risk veterans in community settings.

This application proposes to address this need by evaluating a community-based peer intervention for veterans with opioid use disorder that aims to reduce risk behaviors for opioid-related overdose and HIV/HCV infection. The use of peer-based outreach is designed to reach veteran subpopulations experiencing homelessness, mental health challenges, and significant barriers to healthcare access. Specifically, the intervention to be evaluated will overcome barriers at the three different levels underpinning the theory of triadic influence. Intrapersonal-level barriers for veterans include mental health problems (including PTSD, depression, suicidal ideation), chronic pain, low self-efficacy for behavior change and service involvement, competing priorities related to poverty and homelessness, and distrust of medical systems. Social/interpersonal-level barriers include social isolation, fears of treatment-related stigma (related to military culture), including concerns about the potential impact of seeking treatment on career progression and difficulties interacting with civilians. Last, sociocultural and structural-level barriers, include threats to future career progression represented by a mental health or OUD diagnosis and insufficient education to navigate complex health systems.

The intervention draws on the work of the study team and its experience implementing peer-delivered overdose prevention. This application presents a randomized control trial protocol for assessing a 9-month peer-based intervention employing dedicated veteran specialists to deliver each of the intervention components-education, healthcare/service navigation and social support. These components are all designed to facilitate decreased opioid-related HIV/HCV and OD risk behaviors at the end of the 9-month exposure. The study's specific aims are as follows:

Aim 1: Evaluate the effectiveness of a peer-delivered, community-based education, navigation and support (CENS) intervention to reduce opioid-related risk behaviors (OD/HIV/HCV). The team will use targeted, venue-based sampling to recruit a total of 300 veterans with opioid use disorder. Participants will be randomly assigned (150 each arm) to the 9-month CENS intervention or a 9-month standard naloxone-plus-referrals control and assessed at baseline and at 3-, 6- and 9-months post-baseline, then again at 15-months post-baseline to assess durability of effects. Effectiveness will be measured by treatment and supportive social service utilization and self-reported change in opioid OD52 and HIV/HCV57 risk behaviors.

Aim 2: Examine factors that mediate (e.g., knowledge, self-efficacy, self-stigma) and moderate (e.g., treatment experiences, pain and OUD severity, gender, age) intervention effectiveness.

Aim 3: Explore intervention participants' and peer outreach staff perspectives on implementation as well as barriers to and facilitators of intervention effectiveness. Using in-depth qualitative interviews with a subsample of participants (n=35), service providers (n=10) and peer staff interventionists (n=3), the team will assess participant experiences, psychosocial dynamics underlying intervention effectiveness, and barriers encountered. Findings will be used to inform future implementation and scale-up efforts.

This study stands to contribute a timely, culturally-tailored innovation to overdose prevention-as-usual that, informed by the theory of triadic influence, directly targets the social, intrapersonal, and structural-level barriers to opioid-related risk reduction among veterans. Study findings will be of great interest to community-based and civic healthcare organizations that provide overdose and HIV/HCV risk-reduction outreach, as well as to agencies committed to improving healthcare engagement among veterans.

ELIGIBILITY:
Inclusion Criteria:

* Veteran status
* Adult (18+) age
* Current nonmedical use of opioids
* Current clinical (DSM-5) opioid use disorder of any level of severity

Exclusion Criteria:

* Unable to speak English
* Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Opioid Overdose Risk Behaviors Scale | 9 months follow-up assesment
  Change in Overdose Risk Behavior Scale score, from baseline to 9 months. Min Score= 0 Max Score = 660 Higher scores indicate more engagement in overdose risk behaviors
Change in HIV/HCV Risk Behaviors | 9 months follow-up assessment
  Change in HIV/HCV risk behaviors as measured by the National HIV Behavioral Surveillance System questions about unsafe sexual and injection risk, from baseline to 9 month follow up.

SECONDARY OUTCOMES:
Health service utilization | 9 months follow-up assessment
  Utilization of services as measured by number of visits in past 3 months, e.g. VHA hospitals, syringe exchange, healthcare providers. Measured by the investigator-developed questionnaire.
Drug Treatment | 9 months follow-up assessment
  Utilization of drug treatment in the past 3-months Yes/No Response
HIV/HCV Testing | 9 months follow-up assessment
  Past 3-month number of antibody tests for HIV and HCV

CONTACTS AND LOCATIONS:
Overall Officials: Alexander S Bennett, PhD, Principal Investigator — New York University
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via openICPSR© Self-Deposit Package. All specific identifies will be removed from final datasets prior to release for sharing. To prevent the unlikely but possible deductive disclosure of participant identity with particular characteristics, the study team will make the data available to other investigators only after discussion and under a formal data-sharing agreement that provides for: (1) commitment to use data for research purposes only and not to identify individual study participants; (2) commitment to promote objectivity in research using these data by establishing standards that provide a reasonable expectation that the design, conduct, and reporting of research funded under NIH awards will be free from bias (3) commitment to use appropriate information technology systems to keep data secure; and (4) commitment to returning or destroying data after analyses are complete.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be shared one year after completion of study or by June 2027.
Access Criteria: (1) commitment to use data for research purposes only and not to identify individual study participants; (2) commitment to promote objectivity in research using these data by establishing standards that provide a reasonable expectation that the design, conduct, and reporting of research funded under NIH awards will be free from bias (3) commitment to use appropriate information technology systems to keep data secure; and (4) commitment to returning or destroying data after analyses are complete.